CLINICAL TRIAL: NCT05224336
Title: Behavioral and Neural Mechanisms Supporting Psilocybin-assisted Therapy for Phantom Limb Pain
Brief Title: Psilocybin-assisted Therapy for Phantom Limb Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Fadel Zeidan, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200626
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Phantom Limb Pain
Keywords: Phantom Limb Pain; Psilocybin; Psychedelic Therapy; fMRI; Pain; Chronic Pain; Psychedelics; Hallucinogens; Physiological Effects of Drugs; Psychotropic Drugs
MeSH Terms: conditions — Phantom Limb; Pain; Chronic Pain | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Two sequential studies will be conducted (Study 1 and Study 2). Study 1: The goal of the first study is to assess the feasibility and the corresponding neural mechanisms of administering psilocybin to amputees who are experiencing phantom limb pain. We will perform validated quantitative sensory testing before and after drug administration. Study 1 will have an abbreviated design where participants will receive a single dose of psilocybin (25 mg orally) or placebo (niacin, 100 mg) on one occasion. We will assess psychological, psychophysical pain responses (thermal stimulation) and neural effects before and after administration of psilocybin or placebo.
  Once the first 10 participants complete Study 1, a report documenting their outcomes will be submitted to the UCSD IRB. Once the report is submitted, Study 2 will begin.
  Study 2: The second study will involve two treatment groups; one group will receive psilocybin (25 mg orally) on two occasions, and the second group will receive placeb
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcome assessor will not be made aware if participants are receiving psilocybin or placebo niacin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Participants will receive 25mg oral psilocybin one day to two weeks after baseline psychophysical and fMRI testing. Psychophysical and fMRI testing will then be employed one day to two weeks after drug administration.
  Interventions: Drug: Psilocybin
- Niacin (Placebo Comparator): Participants will receive 100mg oral niacin one day to two weeks after baseline psychophysical and fMRI testing. Psychophysical and fMRI testing will then be employed one day to two weeks after drug administration.
  Interventions: Drug: Placebo Niacin

INTERVENTIONS:
Drug: Psilocybin — 25mg oral psilocybin
  Arms: Psilocybin
Drug: Placebo Niacin — 100mg oral niacin
  Arms: Niacin

SUMMARY:
This double-blind placebo-controlled pilot study seeks to investigate whether psilocybin can be safely administered to people with chronic phantom limb pain (PLP) in a supportive setting with close follow-up, and its effects on pain symptoms and other moods, attitudes, and behaviors. The investigators' primary hypotheses are that psilocybin is safe to administer in people with PLP and that it will reduce scores on measures of pain. The investigators will also assess a number of secondary measures related to the behavioral and neural responses to pain after psilocybin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age
* Amputation of one extremity
* Experience phantom limb pain of at least one month's duration and intensity of at least 3 out of 10 on the VAS
* Able to fluently communicate in English
* Agree to sign the consent and HIPPA authorization
* Willing to refrain from taking serotonergic antidepressant medication during the study period
* Willing to refrain from using any non-prescribed psychoactive drugs, including alcohol, within 24 hours before and after study drug administration
* Agree not to use any nonprescription medications, herbal medications, or supplements during the week prior to each drug session unless an exception is approved by the study investigators
* Willing to refrain from smoking or use of nicotine during the period from 8:00 am on the morning of the drug sessions until they are discharged to go home at the end of the end of the session
* Able to remain in an MRI machine without sedation
* Women of childbearing potential must agree to practice an effective means of birth control throughout the study, from screening to the final visit
* Have a relative or friend who can provide/accompany transportation after the drug session
* If pain is currently being treated with analgesic medications, the analgesic regimen must be stable for at least 2 weeks prior to enrollment, and the participant must agree not to change their use of analgesic medication without first consulting with the study investigators [permissible analgesic medications are as follows: aspirin, acetaminophen, celecoxib, diflunisal, etodolac, fenoprofen, flubiprofen, gabapentin, ibuprofen, indomethacin, ketoprofen, ketorolac, mefenamic acid, meloxicam, nalbumetone, naproxen, pregabalin, proxicam, sulindac, tolmetin, and valdecoxib. PRN use of OTC analgesic medications by participants is also permissible]
* Participants who are taking other medications acting as serotonin antagonists (e.g., cyclobenzaprine, odansetron), dopamine antagonists (e.g., metoclopramide, promethazine, prochlorperazine), dopamine agonists (e.g., levodopa, pramipexole, apomorphine), psychostimulants (e.g., modafinil, armodafinil, solriamfetol, methylphenidate, dexmethylphenidate, atomoxetine, dextroamphetamine, mixed amphetamine salts, lisdexamphetamine), anticholinergics (e.g., benzotropine, trihexyphenidyl, scopolamine, hypscyamine), or N-methyl-D-aspartate receptor antagonists (e.g., amantadine, memantine, ketamine) must be willing to discontinue those medications 1 week prior to each drug session

Exclusion Criteria:

* Under the age of 18 or over the age of 75
* Pregnant or nursing females
* Females of childbearing age who are sexually active but not using birth control
* Phantom limb pain intensity <3 out of 10 on the VAS
* Presence of another type of chronic pain that cannot be differentiated from phantom limb pain by the participant
* Amputation of more than one extremity
* MRI related contraindications including pacemakers, metal implants, spinal cord stimulators etc.
* Meet DSM-V criteria for bipolar disorder, schizophrenia, or other psychotic disorder
* Have a first-degree relative (parent or full-sibling) with a history of bipolar disorder, schizophrenia, or other psychotic disorder
* Judged to present a suicide risk
* Not able to complete an MRI scan
* Active substance use disorder (excluding tobacco and caffeine)
* Subjects prescribed methadone or buprenorphine for any indication
* Require concomitant treatment with efavirenz
* Participants who are prescribed antidepressants or antipsychotics for an axis I diagnosis
* Participants who are taking a serotonergic dietary supplement (e.g., 5-hydroxytryptophan, St. John's wort, SAM-e)
* Participants with any neurological conditions resulting in altered perception or cognition (e.g., dementia, traumatic brain injury, mild cognitive impairment) [with the exception of phantom limb syndrome and its sequelae (depression or anxiety)]
* Participants with a positive urine drug screen for amphetamines, barbiturates, buprenorphine, cocaine, methamphetamine, MDMA, methadone, opiates (morphine, oxycodone), or phencyclidine (PCP)
* Have used psilocybin, psilocybin-containing mushrooms, or another serotonergic hallucinogen (e.g., LSD, mescaline, ayahuasca) for recreational purposes within the last 12 months
* Require concomitant treatment with anti-psychotic medications (aripiprazole, asenapine, brexpiprazole, cariprazine, chlorpromazine, clozapine, fluphenazine, haloperidol, iloperidone, loxapine, mesoridazine, molindone, olanzapine, paliperidone, perphenazine, pimavanserin, pimozide, prochlorpromazine, quetiapine, risperidone, thioridazine, thiothixene, trifluperazine, or ziprasidone)
* Require concomitant treatment with an antidepressant medication or other medications that act as MAO inhibitors or serotonin reuptake inhibitors (amitriptyline, amoxapine, bupropion, citalopram, clomipramine, desipramine, doxepin, duloxetine, escitalopram, fluoxetine, fluvoxamine, imipramine, isocarboxazid, levomilnacipram, maprotiline, milnacipram, mirtazapine, nefazodone, nortriptyline, paroxetine, phenelzine, protriptyline, selegiline, sertraline, tramadol, tranylcypromine, trazodone, trimipramine, venlafaxine, vilazodone, vortioxetine) [trazodone ≤50mg/24hr for insomnia is allowed, but not within 48hr of the psilocybin session]
* Require concomitant treatment with medications known to inhibit UGT1A9 and UGT1A10 (e.g., diclofenac, probenecid, valproic acid)
* Severe hearing or visual impairment
* History of seizure disorder or epilepsy
* History of migraine or other severe recurring headaches necessitating treatment by a neurologist or headache specialist
* History of adverse reactions or intolerance to niacin or the rescue medications used in the study (benzodiazepines, antipsychotics, labetalol, nitroglycerin)
* Presence of uncontrolled cardiovascular disease or uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg)
* Require concomitant treatment with an antihypertensive medication
* QTc prolongation (QTc > 0.045 for man, QTc > 0.047 for women)
* Subjects with history of stroke, angina, clinically significant ECG abnormality (e.g. atrial fibrillation), or artificial heart valve
* Participants with severe renal impairment (GFR < 30 mL/min/1.73 m2)
* Participants with any clinically significant lab abnormalities as determined by a physician on the study team
* Myocardial infarction within the last 12 months
* Participants who meet criteria for Child-Pugh class B or higher
* Participants who are prescribed opioid medications
* Participants taking other medications that may be associated with serotonin syndrome: carbamazepine, dextromethorphan, lithium, linezolid, buspirone
* Evidence of severely compromised hepatic function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Changes in Phantom Limb Pain Intensity | Baseline to Post-Intervention Session (within 2 weeks after session)
  A validated visual analogue scale will be used to quantify the intensity and unpleasantness ratings of phantom limb pain. The minimum rating will be represented as "no pain sensation" or "not at all unpleasant," whereas the maximum was designated with "most intense imaginable" or "most unpleasant imaginable." Higher numbers correspond to higher pain.

SECONDARY OUTCOMES:
Change in Visual Analog Scale Pain ratings | Baseline to Post-Intervention Session (within 2 weeks after session)
  Pain ratings will be assessed in response to the noxious heat stimulation. Pain intensity and unpleasantness ratings will be assessed with a validated visual analog scale. The minimum rating ("0") is labeled as "no pain sensation" or "not at all unpleasant," whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable." Higher numbers correspond to higher pain.
Cerebral Blood Flow (CBF) | Baseline to Post-Intervention Session (within 2 weeks after session)
  Changes in CBF during rest, after intervention session, and during noxious heat stimulation.
Brief Pain Inventory | Baseline to Post-Intervention Session (within 2 weeks after session)
  This is a 7-item self-report measure of pain interference with general activity, mood, walking ability, work, relationships with others, sleep, and enjoyment of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States